CLINICAL TRIAL: NCT01518270
Title: Epidemiologic Analysis of Change in Eyelash Characteristics With Age in Healthy Women
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-LTS-11-003
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Health

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Females: Healthy Females
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment — No treatment will be provided

SUMMARY:
This study will asses epidemiologic changes in eyelash characteristics with increasing age.

ELIGIBILITY:
Inclusion Criteria:

* Willing to have photographs taken of the face/eye regions

Exclusion Criteria:

* No visible eyelashes
* Permanent eyeliner or eyelash implants
* Semi-permanent eyelash tint, dye, or extensions within the last 3 months
* Use of prescription eyelash growth products in the last 6 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Females
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2011-12-16 (Actual); Study Completion 2011-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Irvine, California, United States

REFERENCES:
- [Background] Glaser DA, Jones D, Carruthers J, Campo A, Moench S, Tardie G, Largent J, Caulkins C. Epidemiologic analysis of change in eyelash characteristics with increasing age in a population of healthy women. Dermatol Surg. 2014 Nov;40(11):1208-13. doi: 10.1097/DSS.0000000000000170. PMID 25347452

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Females: Participant's eyelashes were photographed at one study visit.
Period: Overall Study
Arm/Group | Healthy Females
Started | 179
Completed | 179
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Females
Number analyzed (Participants) | 179
Age, Continuous [Mean (Full Range); unit: Years] | 40.3 (10.3) [22.0 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Eyelash Length as Measured by Digital Image Analysis (DIA)
Description: Photographs were taken of the eyelashes. Length was measured in millimeters. Data from both eyes were averaged for each participant for analysis.
Time Frame: Baseline
Population: All participants with values available.
Measure: Mean (Full Range); unit: Millimeters (mm)
Arm/Group | Healthy Females
Number analyzed (Participants) | 177
Millimeters (mm) | 7.33 (1.15) [3.99 to 10.10]

2. Secondary Outcome: Eyelash Thickness as Measured by Digital Image Analysis (DIA)
Description: Photographs were taken of the eyelashes. Eyelash thickness/fullness was assessed across both eyes as an average of the 3 preset areas measured in millimeters squared (mm^2).
Time Frame: Baseline
Population: All participants with values available.
Measure: Mean (Full Range); unit: Millimeters squared (mm^2)
Arm/Group | Healthy Females
Number analyzed (Participants) | 153
Millimeters squared (mm^2) | 1.39 (0.56) [0.32 to 3.13]

3. Secondary Outcome: Eyelash Darkness as Measured by Digital Image Analysis (DIA)
Description: Photographs were taken of the Eyelashes. Eyelash darkness (intensity) was measured within the spline (a narrow area approximately 5 pixels wide that bisects the area of interest). Eyelash darkness was measured in both eyes and averaged for analysis using a scale where 0=black and 255=white.
Time Frame: Baseline
Population: All participants with values available.
Measure: Mean (Full Range); unit: Units on a scale
Arm/Group | Healthy Females
Number analyzed (Participants) | 154
Units on a scale | 122.2 (14.0) [64.7 to 162.5]

ADVERSE EVENTS:
Description: Adverse events were not collected.
Arm/Group | Healthy Females
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.